CLINICAL TRIAL: NCT05783206
Title: Open Multicenter Controlled Clinical Trial to Evaluate Safety and Efficacy of Aerosolized MIR 19 ® Inhalation in Adult Outpatients With Mild COVID-19.
Brief Title: Evaluation of Safety & Efficacy of MIR 19 ® Inhalation Solution in Patients With Mild COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Research Center - Institute of Immunology Federal Medical-Biological Agency of Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-SiCoV/KK46-01/22
Record Dates: First submitted 2023-03-22; First posted 2023-03-24 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: COVID-19; siRNA; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIR 19 ® (Experimental): MIR 19 ® was used in a single dose of 1.85 mg for 3 inhalations per day at intervals of 6-7 hours for 7 days in addition to standard therapy without use of any etiotropic drugs.
  Standard therapy included:
  - paracetamol - 1-2 tablets (500-1000 mg) 2-3 times a day (if body temperature ≥38.0°)
  Interventions: Drug: MIR 19 ®
- Standard therapy (Active Comparator): Standard therapy included:
  * umifenovir (Arbidol®) - 200 mg 4 times per day for 7 days
  * interferon-α, intranasal forms (Grippferon®),spray - in accordance with the instructions.
  * paracetamol - 1-2 tablets (500-1000 mg) 2-3 times a day (if body temperature ≥38.0°)
  Interventions: Combination Product: Standard therapy

INTERVENTIONS:
Drug: MIR 19 ® — MIR 19 ® contains anti-SARS-CoV-2 siRNAs/KK-46 (peptide dendrimer) complexes for inhalation use.
  In the experimental groups treated with MIR 19 ®, the therapy included symptomatic treatment without use of any etiotropic drugs.
  Arms: MIR 19 ®
Combination Product: Standard therapy — Therapy carried out in accordance with the current version of the temporary methodological recommendations of the Ministry of Health of the Russian Federation for the treatment of COVID-19 infection. This therapy included symptomatic treatment as well as etiotropic drugs (except MIR 19 ®)
  Arms: Standard therapy

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of MIR 19 ® in preventing development of moderate and/or severe course of the disease in mild COVID-19 outpatients.

Primary endpoint:

The proportion of patients with the development of moderate or severe COVID-19 disease (in accordance with the criteria specified in the Interim Guidelines "Prevention, diagnosis and treatment of new coronavirus infection (COVID-19)" by the Ministry of Health of the Russian Federation, version 14 of 27.12.2021 or current at the time of the study) by the 28th day of observation.

DETAILED DESCRIPTION:
This is Phase 2b-3 multi-center controlled randomized study to assess the efficacy and safety of MIR 19 ® via 7 days treatment in a dose of 5.55 mg/day of participants with symptomatic mild COVID-19 who did not require hospitalisation.

The MIR 19® is a complex of siRNA, targeting Severe acute respiratory syndrome-related coronavirus 2 (SARS-CoV-2) RNA-dependent RNA polymerase (RdRp) and peptide dendrimer (KK-46).

This study involved 2 cohorts who received:

1. 5.5 mg of the MIR 19 ® per day via inhalation route plus standard therapy which included symptomatic treatment, without any etiotropic drugs.
2. Standard therapy which included symptomatic treatment as well as etiotropic drugs except MIR 19 ®.

All subjects will undergo scheduled safety and efficacy assessments as outpatients to the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18 who have been diagnosed with COVID-19 and who need therapy on an outpatient basis according to the Interim Guidelines "Prevention, diagnosis and treatment of new coronavirus infection (COVID-19)"by Ministry of Health of the Russian Federation. Version 14 from 12/27/2021.
* Able to give informed consent and attend all study visits
* Duration of the disease from the first symptoms (presence of at least one of the following symptoms: fever, cough, myalgia, weakness, shortness of breath, headache, nausea, stool disorders, loss of appetite) up to the day of screening no more than 5 days.
* Negative pregnancy test for women with preserved reproductive potential
* Participants must agree to use the reliable contraception while on study medication and for posttrial contraception for 3 month
* The patient's ability to inhale the experimental drug

Exclusion Criteria:

* Respiratory rate is more than 22 / min
* Oxygen saturation - SpO2 ≤ 94%.
* Decreased level of consciousness, agitation.
* Unstable hemodynamics (systolic blood pressure less than 100 mmHg or diastolic blood pressure less than 60 mmHg).
* Long-term systemic corticosteroid exposure.
* Autoimmune or inflammatory diseases (systemic / localized), as well as oncological diseases.
* Symptoms of moderate, severe or critical COVID-19 at the time of screening
* Positive blood tests for HIV, hepatitis B and С, syphilis.
* Pregnancy and breast-feeding.
* Previous adverse reactions to the active substance and/or excipients included in the drug
* Chronic diseases of the cardiovascular system
* Type 1 diabetes.
* The following laboratory parameters are excluded: Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, total and direct bilirubin >4 x upper limit of normal (ULN);
* C-reactive protein (CRP) level > 10 mg/L.
* Participation in other investigational drug or device clinical trials within 90 days prior to screening.
* History of alcohol, drug or chemical abuse
* Previous hospitalizations associated with the development of moderate and severe COVID-19.
* Mental illness.
* Receipt of plasma from a person who recovered from COVID-19 (convalescent plasma) up to 14 days before participating in the study, vaccination against SARS-CoV-2 less than 4 weeks before randomization.
* Any conditions that, according to the researcher's, may be a contraindication to the participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Moderate or severe COVID-19 | 28th day of observation
  The proportion of patients with the development of moderate or severe COVID-19 disease (in accordance with the criteria specified in the Interim Guidelines "Prevention, diagnosis and treatment of new coronavirus infection (COVID-19)" by the Ministry of Health of the Russian Federation, version 14 of 27.12.2021 or current at the time of the study)

SECONDARY OUTCOMES:
Etiotropic therapy | 28th day of observation
  The proportion of patients required another etiotropic therapy COVID-19 during the study.
Severity of COVID-19 symptoms | 28th day of observation
  Assessment of the severity of COVID-19 symptoms (nasal congestion, sore throat, shortness of breath, cough, weakness, myalgia, headache, chills, fever, nausea, vomiting, diarrhea, anosmia, ageusia) according to the patient's diary.
Results of polymerase chain reaction (PCR) | 28th day of observation
  The proportion of patients with negative PCR to SARS-CoV-2 at visits 4, 5
Improvement / disappearance of COVID-19 symptoms | 28th day of observation
  Time to clinical improvement / disappearance of symptoms according to the scale of assessment of the severity of symptoms of the disease
Duration of COVID-19 symptoms | 28th day of observation
  Duration of clinical symptoms of COVID-19 disease (fever, cough, myalgia, weakness, shortness of breath, headache, nausea, stool disorders, loss of appetite, anosmia, ageusia) according to the patient's diary.
Moderate COVID-19 | 28th day of observation
  Proportion of patients with moderate COVID-19.
Severe COVID-19 | 28th day of observation
  Proportion of patients with severe COVID-19.
Critical COVID-19 | 28th day of observation
  Proportion of patients with critical COVID-19
Hospitalization | 28th day of observation
  Proportion of hospitalized patients
Death rate | 28th day of observation
  The proportion of deaths during the study
Worsening of COVID-19 symptoms | 28th day of observation
  The proportion of patients with worsening of COVID-19 clinical symptoms during the study by at least 1 point

CONTACTS AND LOCATIONS:
Locations (1):
- NRC Institute of Immunology FMBA, Moscow, Russia